CLINICAL TRIAL: NCT02949518
Title: Enhanced Recovery After Spine Surgery: A Prospective Randomized Controlled Trial to Assess Quality of Recovery and the Biochemical Stress Response to Lumbar Fusion
Brief Title: Enhanced Recovery After Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2016-617
Record Dates: First submitted 2016-10-07; First posted 2016-10-31 (Estimated); Results first posted 2020-07-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Enhanced Recovery After Surgery; Spine Surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Enhanced Recovery Pathway for Spine (Experimental)
  Interventions: Other: Enhanced Recovery Pathway (ERP) for Spine
- Usual Care (No Intervention)

INTERVENTIONS:
Other: Enhanced Recovery Pathway (ERP) for Spine — The study team emphasizes that all components of the ERP are considered standard of care at this institution. The objective of this study is to ensure that the study patients assigned to the ERP will receive these standard of care components.
  Arms: Enhanced Recovery Pathway for Spine

SUMMARY:
Enhanced recovery pathways (ERP) after surgery have been shown to decrease length of stay and perioperative complications in a range of surgical specialties. To date, ERPs has not been studied in patients presenting for spine surgery. The investigators have recently developed an interdisciplinary pathway for spine surgery patients based on the latest available evidence and guidelines. The aim of this trial is to compare the investigators enhanced recovery pathway with conventional perioperative management in patients undergoing 1-2 level posterior lumbar fusion.

ELIGIBILITY:
Inclusion Criteria:

* Any patient presenting for 1 or 2 level posterior lumbar fusion.

Exclusion Criteria:

* Cognitive impairment (baseline dementia, cognitive dysfunction or inability to consent to participate).
* Kidney disease: GFR <60 mL/min/1.73 m2 for 3 months or more, irrespective of cause (Levey et al., 2012).
* Liver disease: transaminitis, cirrhosis, hepatitis, hypoalbuminemia, coagulopathy.
* Pre-existing bowel disease (inflammatory bowel disease, colectomy/ colostomy/diverticular disease).
* Allergy/intolerance/contraindication to any medication or component included in the ERAS pathway protocol.
* Patients whose primary or preferred language is not English.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Soffin, MD, PhD, Principal Investigator — Hospital for Special Surgery, NY
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Enhanced Recovery Pathway: An evidence-based enhanced recovery pathway for 1- and 2-level open lumbar fusion based on Enhanced Recovery After Surgery™ Society principles of care. The study team emphasizes that all components of the ERAS pathway are considered standard of care at this institution.
- Usual Care: Anesthesiologist/surgeon in charge of patients randomized to the usual care arm had sole discretion over intraoperative treatment and there were no specific study interventions.
Period: Overall Study
Arm/Group | Enhanced Recovery Pathway | Usual Care
Started | 28 | 28
Completed | 25 | 26
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Recovery Pathway | Usual Care | Total
Number analyzed (Participants) | 25 | 26 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (18.1) | 54.2 (13.7) | 54.5 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 18 | 29
  Male | 14 | 8 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 25 | 24 | 49
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 24 | 22 | 46
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
ASA Level [Count of Participants; unit: Participants] — ASA 1: A normal healthy patient. ASA 2: A patient with a mild systemic disease. ASA 3: A patient with a severe systemic disease that is not life-threatening.
  Participants
    ASA I | 6 | 6 | 12
    ASA II | 18 | 19 | 37
    ASA III | 1 | 1 | 2
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.1 (4.2) | 29.4 (5.3) | 28.26 (4.89)
Total Anesthesia Time [Mean (Standard Deviation); unit: minutes] | 269 (57) | 268.5 (63.8) | 268.76 (59.91)
Total Surgery Time [Mean (Standard Deviation); unit: minutes] | 183.2 (54) | 192.3 (62.4) | 187.84 (58.0)
Surgery Fusion Level [Count of Participants; unit: Participants] — Type of Surgery - either 1 Level or 2 Level Spine Fusion was done.
  Fusion of only one motion segment of the spine (e.g. L5-S1) is referred to as a 1 level fusion. 2-level fusion may be considered for patients with severe, disabling pain that occurs at two levels of the spine (e.g. L4-L5 and L5-S1).
  Participants
    Fusion Level I | 21 | 21 | 42
    Fusion Level II | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Patient Score on QoR40 Inventory.
Description: The Quality of Recovery 40 (QoR40) is a 40-item questionnaire which assesses five dimensions of recovery after surgery and anesthesia: comfort, emotions, physical independence, patient support and pain. The QoR40 has been validated for both clinical and research use. The QoR-40 has a possible score of 40 (extremely poor quality of recovery) to 200 (excellent quality of recovery).
Time Frame: Postoperative Day 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Enhanced Recovery Pathway (ERP) for Spine: he study team emphasizes that all components of the ERP are considered standard of care at this institution. The objective of this study is to ensure that the study patients assigned to the ERP will receive these standard of care components.
- Usual Care: anesthesiologist/surgeon in charge of patients randomized to the usual care arm had sole discretion over intraoperative treatment
Arm/Group | Enhanced Recovery Pathway (ERP) for Spine | Usual Care
Number analyzed (Participants) | 22 | 25
scores on a scale | 179.4 (13.79) | 170.3 (15.49)

2. Secondary Outcome: Length of Stay and Time From Surgery to Meeting Discharge and Physical Therapy Goals.
Description: Measured in days after surgery (in half-day increments).
Time Frame: Postoperative Day 5
Population: One patient did not meet physical therapy goals
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Enhanced Recovery Pathway | Usual Care
Number analyzed (Participants) | 25 | 26
days
  Length of Stay | 2.8 [2.1 to 3.7] | 3.1 [2.8 to 4.8]
  Time to meet physical therapy goals: number analyzed (Participants) | 24 | 26
  Time to meet physical therapy goals | 1.4 [1 to 2.4] | 1.9 [1.8 to 2.9]

3. Secondary Outcome: Pain Control: Opioid Consumption.
Description: Measured in morphine equivalents daily.
Time Frame: 48 hours after surgery
Population: Patients who were discharged between the 24-48 hour time mark did not have data collected.
Measure: Median (Inter-Quartile Range); unit: morphine equivalents daily
Arm/Group | Enhanced Recovery Pathway | Usual Care
Number analyzed (Participants) | 24 | 26
morphine equivalents daily
  0-24 Hours | 61.8 [25.6 to 103.3] | 133.2 [39.5 to 218.3]
  24-48 Hours: number analyzed (Participants) | 18 | 25
  24-48 Hours | 30 [20 to 97.5] | 75 [28 to 120]

4. Secondary Outcome: Pain Control: NRS Rating Scales of Pain After Physical Therapy on Postoperative Day 1
Description: Scale of 0-10, 0 being no pain, 10 being the worst pain possible
Time Frame: Postoperative Day 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Enhanced Recovery Pathway | Usual Care
Number analyzed (Participants) | 24 | 23
units on a scale | 3 [0.5 to 3] | 4 [3 to 5]

5. Secondary Outcome: Time to Post-operative Oral Intake.
Description: Measured in hours
Time Frame: Postoperative Day 1
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Enhanced Recovery Pathway | Usual Care
Number analyzed (Participants) | 25 | 26
hours | 5.1 [2.9 to 7.7] | 7.9 [5.5 to 13.5]

6. Secondary Outcome: Number of Participants With Post-operative Nausea, Vomiting and Ileus
Description: If the patient ever had any of the events of nausea, vomiting, ileus by day of discharge
Time Frame: Postoperative Day 5
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Recovery Pathway | Usual Care
Number analyzed (Participants) | 25 | 26
Participants
  Nasea | 8 | 13
  Vomiting | 3 | 2
  Ileus | 4 | 6

7. Secondary Outcome: Levels of Plasma Markers of Surgical Stress: IL-6 (pg/ml).
Time Frame: Postoperative Days 0, 1, and 3
Population: Patients who were discharged before Postoperative Day 3 did not have data collected.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Enhanced Recovery Pathway | Usual Care
Number analyzed (Participants) | 25 | 25
pg/mL
  Postoperative Day 0 | 2.5 [2.5 to 5] | 2.5 [2.5 to 5]
  Postoperative Day 1 | 5 [2.5 to 7] | 5 [2.5 to 8]
  Postoperative Day 3: number analyzed (Participants) | 14 | 22
  Postoperative Day 3 | 8 [6 to 19] | 8 [6 to 21]

8. Secondary Outcome: Levels of Plasma Markers of Surgical Stress: Cortisol (mcg/dl).
Time Frame: Postoperative Days 0, 1, and 3
Population: Patients who were discharged before Postoperative Day 3 did not have data collected.
Measure: Median (Inter-Quartile Range); unit: mcg/dl
Arm/Group | Enhanced Recovery Pathway | Usual Care
Number analyzed (Participants) | 25 | 26
mcg/dl
  Postoperative Day 0 | 6.3 [2.4 to 7.9] | 5.4 [2.2 to 14]
  Postoperative Day 1 | 0.5 [0.5 to 0.5] | 0.5 [0.5 to 1.5]
  Postoperative Day 3: number analyzed (Participants) | 14 | 22
  Postoperative Day 3 | 8.3 [3.1 to 10.6] | 8.9 [6.9 to 13.9]

9. Secondary Outcome: Levels of Plasma Markers of Surgical Stress: CRP (mg/dL).
Time Frame: Postoperative Days 0, 1, and 3
Population: Patients discharged before postoperative day 3 did not have data collected.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Enhanced Recovery Pathway | Usual Care
Number analyzed (Participants) | 25 | 26
mg/dL
  Postoperative Day 0 | 0.4 [0.4 to 0.7] | 0.4 [0.4 to 0.7]
  Postoperative Day 1 | 1.6 [0.9 to 2.5] | 1.6 [1.1 to 2.2]
  Postoperative Day 3: number analyzed (Participants) | 14 | 22
  Postoperative Day 3 | 6.1 [3.8 to 15.7] | 15.9 [6.6 to 19.7]

10. Secondary Outcome: Levels of Plasma Markers of Surgical Stress: Insulin Resistance (µIU/ml).
Time Frame: Postoperative Days 0, 1, and 3
Population: Patients discharged before postoperative day 3 did not have data collected.
Measure: Median (Inter-Quartile Range); unit: uIU/mL
Arm/Group | Enhanced Recovery Pathway | Usual Care
Number analyzed (Participants) | 25 | 25
uIU/mL
  Postoperative Day 0 | 8 [5 to 11] | 10 [7 to 15]
  Postoperative Day 1 | 15 [10 to 28] | 14 [8 to 20]
  Postoperative Day 3: number analyzed (Participants) | 14 | 22
  Postoperative Day 3 | 18 [13 to 46] | 15.5 [6 to 26]

11. Secondary Outcome: Number of Participants With Presence of Delirium/Confusion, Infection, DVT/PE
Description: Incidence of patients with event of delirium/confusion, infection, DVT/PE will be assessed for the entire hospital admission but measured at discharge.
Time Frame: Entire Hospital Admission, but Measure at Discharge (Up to Postoperative Day 5)
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Recovery Pathway | Usual Care
Number analyzed (Participants) | 25 | 26
Participants
  Delirium/Confusion | 1 | 2
  Infection | 1 | 0
  DVT/PE | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected during their length of stay in the hospital (which as at most up to 5 days) after surgery.
Description: The risks of collecting plasma for this study are similar to the risks of a routine blood draw, including - mild pain, bruising, and very rarely infection at the place of needle insertion. However, the likelihood of these risks occurring is rare, as an arterial line catheter is routinely placed in patients undergoing this class of spine surgery in order to continuously monitor the patient's hemodynamics perioperatively. The study team expected to draw samples using the pre-existing catheter.
Arm/Group | Enhanced Recovery Pathway | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/26
Other Adverse Events (participants affected / at risk) | 0/25 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/18/NCT02949518/Prot_SAP_000.pdf